CLINICAL TRIAL: NCT03813368
Title: Short and Long Term Outcomes of Whipples Resection in the Over 80s
Brief Title: Whipples Resection in Octogenarians
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 258426
Record Dates: First submitted 2018-12-10; First posted 2019-01-23 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Whipples pancreatico-duodenectomy — Classic whipples and pylorus preserving

SUMMARY:
Whipples resection is an operation that has a burden of high morbidity and mortality. It is performed for a variety of disorders of the pancreas, duodenum and ampulla. The most common indication is pancreatic ductal adenocarcinoma which has a poor long term outcome even when curative surgery has been performed. Short and long term outcomes however, have improved recently and the indications for curative resection have been increasingly extended, including operating on those that previously may have been considered too old to benefit from curative resection.

Little is known about the benefit of performing this procedure in the oldest patients. Performing Whipples resection in patients over the age of 70 has been reported and has been shown to result in satisfactory perioperative results with comparable long term outcomes to those under 70. However the benefit of performing the same procedure in the over 80 age group is less well reported and consistently presents a challenging decision for the clinician.

DETAILED DESCRIPTION:
Whipples resection is an operation that has a burden of high morbidity and mortality. It is performed for a variety of disorders of the pancreas, duodenum and ampulla. The most common indication is pancreatic ductal adenocarcinoma which has a poor long term outcome even when curative surgery has been performed. Short and long term outcomes however, have improved recently and the indications for curative resection have been increasingly extended, including operating on those that previously may have been considered too old to benefit from curative resection.

Little is known about the benefit of performing this procedure in the oldest patients. Performing Whipples resection in patients over the age of 70 has been reported and has been shown to result in satisfactory perioperative results with comparable long term outcomes to those under 70. However the benefit of performing the same procedure in the over 80 age group is less well reported and consistently presents a challenging decision for the clinician.

This study therefore aims to assess the short and long term outcomes of patients undergoing Whipples PD in the over 80 age group in Lothian. This will be combined with data from all the other units in Scotland that perform Whipples resection (Dundee, Glasgow and Aberdeen)

The primary outcome will be overall and disease free survival.

Participants will be identified by using procedure specific codes to identify those patients who underwent Whipples pancreaticoduodenectomy from the ORSOS prospectively collated theatre record database. The other centres in Scotland will identify their subjects via their own methodology.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing Whipples PD from 1998-2018 in Scotland

Exclusion Criteria:

* incorrectly coded as Whipples resection
* Underwent non curative bypass procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had whipples pancreatico-duodenectomy in Scotland
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
survival | 10 years
  Time from surgery to death
Disease free survival | 10 years
  Time from surgery to recurrence

SECONDARY OUTCOMES:
Morbidity | 90 days
  Clavien Dindo grade of post-oepraitve complication
Discharge Destination | 5 years
  Where the patient has been discharged from hospital to - home, nursing home, care home, home with support

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hughes, Principal Investigator — NHS Lothian
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided